CLINICAL TRIAL: NCT02950103
Title: Efficacy and Safety Evaluation of Synthetic Phosphoethanolamine in Solid Tumor Patients
Brief Title: Efficacy and Safety of Synthetic Phosphoethanolamine in Solid Tumor Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Secretaria de Estado da Saúde (Other Government)
Collaborators: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP977
Record Dates: First submitted 2016-09-26; First posted 2016-10-31 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Solid Tumor
Keywords: solid tumor; phase II; phosphoethanolamine
MeSH Terms: interventions — phosphorylethanolamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Synthetic phosphoethalonamine (Experimental): Phosphoethanolamine PO daily
  Interventions: Drug: Phosphoethanolamine

INTERVENTIONS:
Drug: Phosphoethanolamine — Phosphoethanolamine PO daily

SUMMARY:
Synthetic phosphoethanolamine is a primary amine which has a critical role in the biosynthesis of cell membranes. Pre-clinical models have shown potential anticancer activity.

DETAILED DESCRIPTION:
Phase II multi-cohort study based on two-stage Simon design. The primary goal of the study is response rate at 8 weeks in participants with advanced solid tumors treated with synthetic phosphoethanolamine, as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1) or specific criteria for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven advanced solid tumor patients (recurrent or metastatic), not amenable to curative therapy. Patients must have progressed to standard treatment proven to prolong survival or no standard treatment exists. Tumor types include head and neck squamous cell carcinoma, non-small cell lung cancer, colorectal adenocarcinoma, breast cancer, cervix cancer, prostate cancer, melanoma, pancreas adenocarcinoma, gastric adenocarcinoma, hepatocellular carcinoma
* No concurrent active systemic treatment
* Measurable disease by RECIST v1.1
* Clinical or radiological progression in the last three months
* Eastern Cooperative Oncology Group Performance Status 0-1
* Ability to consent
* Adequate organ function
* Life expectancy greater than 12 weeks
* Ability to swallow
* No previous malignancy in the last 5 years

Exclusion Criteria:

* Pregnancy
* Corticosteroid therapy for prostate cancer
* Uncontrolled comorbidity
* Known hepatitis B, C and HIV
* Central nervous system involvement, except if controlled symptoms and without corticosteroids
* Previous use of phosphoethalonamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-08; Primary Completion 2017-03 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
RECIST v 1.1 response rate or specific criteria for prostate cancer | 8 weeks

SECONDARY OUTCOMES:
Treatment related toxicities as determined by CTCAE version 4.0 | Every cycle, up to 30 days after drug interruption
Overall survival | Survival followed every 2 months from inclusion until death, withdrawal, loss to follow-up, or study end for up to 60 months
Disease free survival | Tumor assessment by RECIST v1.1 or prostate cancer specific criteria every 8 weeks for up to 12 months, then every 12 weeks until loss of clinical benefit, withdrawal, death, or study end for up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No